CLINICAL TRIAL: NCT03247868
Title: Multimodal Treatment of Cervical Dystonia With Botulinum Toxin Injections Associated With a Sensory-motor Perceptive Rehabilitation Integrated Approach (SPRInt) Based on Motor Learning Techniques
Brief Title: A Multimodal Approach to Cervical Dystonia Treatment With Association of Botulinum Toxin and Motor Learning Techniques
Acronym: SPRInt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SPRIntFdG
Record Dates: First submitted 2017-07-27; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Cervical Dystonia,Primary
MeSH Terms: conditions — Cervical Dystonia, Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Botulinum toxin+SPRInt protocol (Experimental): patients affected by cervical dystonia receive botulinum toxin treatment (EMG-US guided injections in dystonic muscles) for two times at T0 and T2; after T2 patients are treated also with SPRInt rehabilitation protocol based on motor learning techniques.
  Interventions: Combination Product: Botulinum Toxin+SPRInt

INTERVENTIONS:
Combination Product: Botulinum Toxin+SPRInt — Botulinum toxin injections in association with rehabilitative approach to cervical dystonia (SPRInt)

SUMMARY:
the aim of this study protocol is to describe, using a longitudinal study, a multimodal approach of treatment of cervical dystonia with botulinum toxin (BoNTA) and a new rehabilitation protocol named SPRInt (Sensory-motor perceptive rehabilitation integrated) approach based on motor learning techniques and spatial rehabilitation.

DETAILED DESCRIPTION:
Longitudinal study utilizing a multimodal treatment protocol developing in six months time:

Phase 1 : BoNTA injections localized in dystonic cervical muscles with EMG/US guides performed after polygraphy and kinematic analysis of cervical region Times: T0: pre treatment; T1: 6 weeks after T0 considered BoNTA pharmacological peak effect; T2: 12 weeks after T0 considered from guidelines and pharmaceutical data sheet the lowest BoNTA effect.

Phase 2: BoNTA performed in the same way of Phase 1 associated to SPRInt protocol Times: T2: before combination of BoNTA and rehabilitation treatment (18 sessions of 45 minutes three times a week); T3: 6 weeks after T2 considered BoNTA pharmacological peak effect and the end of SPRInt protocol; T4: 12 weeks after T2 considered from guidelines and pharmaceutical data sheet the lowest BoNTA effect and follow up of SPRInt-consolidation.

The SPRInt approach aims are to improve body perception, posture and movement quality and to restore body axis by using specific sensory feedbacks, both intrinsic (IFB) and extrinsic (EFB), and motor exercises (ME) with specific rhythmic temporal structure.The ME can be focused on different body parts (eyes, head, neck, trunk, arm) and involve different spatial planes (frontal, sagittal, horizontal, multiplanar).

The exercises can be performed with eyes closed and with an external passive motor leading in order to improve proprioception and facilitate sensory integration by excluding visual or verbal information that can be misleading for the patient. The ability to perceive and integrate intrinsic feedback is the fundamental element to create mental image that define body scheme and motor behaviour.

The extrinsic feedback can be continuous or discontinuous (on-off timing) and gives the patient information about the performance or result by positive or negative reinforcement; this process can be important to motivate and empower the patient in reaching new skills.

The final goal for the patient is to reinforce and retain the informations collected with working memory and then stored with the consolidation process which ends in learning new skills (ie rescue postural axis) and improving motor tasks (ie move the head in the opposite position).

At each time point these test are performed:

* CLINICAL SCALES i. Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS)

  1. Severity
  2. Disability
  3. Pain ii. Quality of life iii. Depression Beck Scale iv. Zung Self Rating Anxiety Scale v. Rey Test to test visuo spatial abilities
* MOVEMENT ANALYSIS and KINEMATIC AND EMG MAPPING of cervical region ( head and neck)
* FUNCTIONAL MAGNETIC RESONANCE BRAIN STUDY to perform brain measurements of functional connectivity (resting state-Default Mode Network), morphometry (volume, area, cortical thickness, cortical curvature, node degree) and tractography.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 yo
* diagnosis of idiopathic cervical dystonia
* disease duration more than 6 months

Exclusion Criteria:

* diagnosis of secondary dystonia on previously performed neuroimaging data (ie structural lesion of cervical spine, vascular or traumatic brain injuries)
* history of neuroleptic drug treatment (antidopaminergic drugs)
* associated neurological illness
* botulinum toxin treatment in the 3 previous months before recruitment
* head tremor without dystonic posturing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-03-16; Primary Completion 2018-03-28 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Dystonia phenomenology improvement | every six weeks during six months time
  a clinical assessment of dystonia will be conducted at each study visit using TWSTRS

SECONDARY OUTCOMES:
quality of life | every six weeks during six months time
  a clinical assessment of dystonia severity will be conducted at each study visit using quality of life scale (EQ5D5L)
brain plasticity | every six weeks during six months time
  study of functional connectivity using functional magnetic resonance
depression | every six weeks during six months time
  depression scale (BECK)
anxiety | every six weeks during six months time
  anxiety scale (ZUNG)
structural grey matter plasticity | every six weeks during six months time
  brain study of morphometry using functional magnetic resonance
structural white matter plasticity | every six weeks during six months time
  tractography of brain areas using functional magnetic resonance
kinematic assessment of dystonia severity | every six weeks during six months time
  visit with optoelectronic system

CONTACTS AND LOCATIONS:
Overall Officials: Anna Castagna, MD, Principal Investigator — IRCCS Fondazione Don Gnocchi
Locations (1):
- IRCCS Fondazione Don Gnocchi, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Albanese A, Bhatia K, Bressman SB, Delong MR, Fahn S, Fung VS, Hallett M, Jankovic J, Jinnah HA, Klein C, Lang AE, Mink JW, Teller JK. Phenomenology and classification of dystonia: a consensus update. Mov Disord. 2013 Jun 15;28(7):863-73. doi: 10.1002/mds.25475. Epub 2013 May 6. PMID 23649720
- [Background] Boccagni C, Carpaneto J, Micera S, Bagnato S, Galardi G. Motion analysis in cervical dystonia. Neurol Sci. 2008 Dec;29(6):375-81. doi: 10.1007/s10072-008-1033-z. Epub 2008 Nov 29. PMID 19043661
- [Background] Walter U, Dressler D. Ultrasound-guided botulinum toxin injections in neurology: technique, indications and future perspectives. Expert Rev Neurother. 2014 Aug;14(8):923-36. doi: 10.1586/14737175.2014.936387. Epub 2014 Jul 21. PMID 25046267
- [Background] Prudente CN, Hess EJ, Jinnah HA. Dystonia as a network disorder: what is the role of the cerebellum? Neuroscience. 2014 Feb 28;260:23-35. doi: 10.1016/j.neuroscience.2013.11.062. Epub 2013 Dec 11. PMID 24333801
- [Background] Delnooz CC, Pasman JW, van de Warrenburg BP. Dynamic cortical gray matter volume changes after botulinum toxin in cervical dystonia. Neurobiol Dis. 2015 Jan;73:327-33. doi: 10.1016/j.nbd.2014.10.013. Epub 2014 Oct 28. PMID 25447226
- [Background] Delnooz CC, Pasman JW, Beckmann CF, van de Warrenburg BP. Task-free functional MRI in cervical dystonia reveals multi-network changes that partially normalize with botulinum toxin. PLoS One. 2013 May 1;8(5):e62877. doi: 10.1371/journal.pone.0062877. Print 2013. PMID 23650536
- [Background] De Pauw J, Van der Velden K, Meirte J, Van Daele U, Truijen S, Cras P, Mercelis R, De Hertogh W. The effectiveness of physiotherapy for cervical dystonia: a systematic literature review. J Neurol. 2014 Oct;261(10):1857-65. doi: 10.1007/s00415-013-7220-8. Epub 2014 Jan 12. PMID 24413637
- [Background] van den Dool J, Visser B, Koelman JH, Engelbert RH, Tijssen MA. Cervical dystonia: effectiveness of a standardized physical therapy program; study design and protocol of a single blind randomized controlled trial. BMC Neurol. 2013 Jul 15;13:85. doi: 10.1186/1471-2377-13-85. PMID 23855591
- [Background] Simpson DM, Hallett M, Ashman EJ, Comella CL, Green MW, Gronseth GS, Armstrong MJ, Gloss D, Potrebic S, Jankovic J, Karp BP, Naumann M, So YT, Yablon SA. Practice guideline update summary: Botulinum neurotoxin for the treatment of blepharospasm, cervical dystonia, adult spasticity, and headache [RETIRED]: Report of the Guideline Development Subcommittee of the American Academy of Neurology. Neurology. 2016 May 10;86(19):1818-26. doi: 10.1212/WNL.0000000000002560. Epub 2016 Apr 18. PMID 27164716
- [Background] Curra A, Trompetto C, Abbruzzese G, Berardelli A. Central effects of botulinum toxin type A: evidence and supposition. Mov Disord. 2004 Mar;19 Suppl 8:S60-4. doi: 10.1002/mds.20011. PMID 15027056
- [Background] Kitago T, Krakauer JW. Motor learning principles for neurorehabilitation. Handb Clin Neurol. 2013;110:93-103. doi: 10.1016/B978-0-444-52901-5.00008-3. PMID 23312633
- [Derived] Castagna A, Caronni A, Crippa A, Sciume L, Giacobbi G, Corrini C, Montesano A, Ramella M. Sensorimotor Perceptive Rehabilitation Integrated (SPRInt) program: exercises with augmented movement feedback associated to botulinum neurotoxin in idiopathic cervical dystonia-an observational study. Neurol Sci. 2020 Jan;41(1):131-138. doi: 10.1007/s10072-019-04061-5. Epub 2019 Sep 2. PMID 31478151